CLINICAL TRIAL: NCT03281447
Title: NaviCan. Navigation and Support to Cancer Patients - A Randomized Controlled Trial.
Brief Title: Nurse Navigation Versus Current Care Coordination During Colorectal Cancer Trajectories
Acronym: NaviCan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); Laval University (Other); Slagelse Hospital (Other); Region of Southern Denmark (Other); Region Zealand (Other); Danish Cancer Society (Other); Odense Patient Data Explorative Network (Other)
Responsible Party: Principal Investigator, Marianne K. Thygesen, Associate professor, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 020-2016-NQ; 2008-58-0035 (Other: the Danish Data Protection Agency)
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Self Efficacy; Continuity of Care; Quality of Life; Colorectal Neoplasms; Case Management
Keywords: Nurse navigation; Family; Self Efficacy; Needs assessment; Quality of Life; Colorectal Neoplasms; Case Management
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nurse navigation (Experimental): Coherent navigation and support from a family-centred viewpoint throughout the cancer trajectory, despite the individual patient's affiliation to any department.
  Interventions: Other: Nurse navigation
- Current care coordination (Active Comparator): Department-specific coordination and answers to questions from a patient-centred viewpoint.
  Interventions: Other: Current care coordination

INTERVENTIONS:
Other: Nurse navigation
  Arms: Nurse navigation
Other: Current care coordination
  Arms: Current care coordination

SUMMARY:
In western countries, the number of cancer survivors increases, and current cancer care seems insufficient with both patients' experiences of lack of help in transitions and up to 60 % of the patients having psychological problems after treatment. Further, Denmark shall have new hospitals, where researchers and healthcare professionals are expected to merge tasks and reach a higher patient experienced quality of care, without additional costs, so a better way to provide cancer care, which benefits the patients and supports the ideas within the new hospitals in Denmark, is needed.

In a randomized controlled trial, the organizational structure of the healthcare system is challenged and the impact of a coherent nurse navigation practice compared to the currently existing department-specific care coordination is tested. The primary data are changes in patients' self-reported cancer-related self-efficacy from inclusion till one week after receipt of the information that they have reached the end of treatment, or in case of prolonged treatment, till not later than one year after inclusion.

Patients can participate if they are 18 years of age or older, speak and understand Danish, and have a proven lesion suspected of cancer in the colon or rectum after colonoscopy or sigmoidoscopy at the Danish endoscopy centers at Odense University Hospital (the cities: Nyborg, Svendborg and Odense) or at Slagelse Hospital. Furthermore, participants must not be mentally retarded, they must not suffer from a constant life-threatening disease, and they must not suffer from, or be in the diagnostic phase of, dementia or severe psychiatric disease.

Participants are allocated to support from nurse navigation or to current care coordination, and fill in four questionnaires during their cancer trajectory: 1) At inclusion, 2) Three days before treatment start, 3) One week after receipt of information about treatment end or not later than one year after inclusion, and 4) Six weeks after measure point 3. Data is analyzed using suitable statistical models.

With positive results, participants in nurse navigation are better helped during their cancer trajectory and have a better psychological start on the rest of their lives after cancer treatment. Focus will be on colon and rectum cancer care, but the results will be transferable to similar settings. Furthermore, positive results will support changes in the onset of rehabilitation initiatives.

DETAILED DESCRIPTION:
The primary hypothesis in this study is:

Nurse navigation, as a specific, defined concept of coherent help through cancer trajectories, will prove superior to current care coordination with regard to patients' self-evaluated self-efficacy for cancer from inclusion to one week after receipt of information about treatment end or not later than one year after inclusion.

Allocation The randomization will be stratified by age and gender. The rational is that age and gender is differently associated with benefit by a given care.

Data collection Participants fill in questionnaires at four measurements, and supplements to sociodemographic information as well as information for an economic evaluation is collected from provider side.

The questionnaires for participants are available in paper and electronically, and participants are allowed to discuss the individual questions with a person whom they trust before filling in their answers. If a participant is blind or dyslexic and has no one to help them fill in the questionnaires, a trained study nurse will read out loud the questions and fill in the participant's answers, and eventually in this process, listen to the participant's pros and cons, acknowledge that they are heard, ask for an answer and read out loud the question again. All data are stored in Research Electronic Data Capture (RedCap).

Blinding The trial is not blinded but all participants are told, there is no favorite group. The statistician is blinded to randomization group and this blinding will be unveiled after the data is analyzed.

Statistics Data are analyzed following the modified intention-to-treat principle, which is carried out by a senior statistician in close collaboration with the research group. Usual descriptive statistics will be used to summarize baseline and subject characteristics. The analyses of the primary endpoint, i.e. change in self-evaluated self-efficacy for cancer from inclusion (measurement 1) to end of treatment (measurement 3), and the secondary outcomes are done using analysis of covariance of the measure at measurement 3 with randomization group as a factor and measure at measurement 1 as covariate. In secondary analyses for all endpoints (measurement 1-4), the change over time will be investigated by mixed effects repeated measures analysis with randomization group as factor and random effects for subjects. These analyses are repeated within the subgroup of all cancer patients and the subgroup of cancer patients treated with curative aim. In the subgroup analyses, the influence of relevant subject-level confounders such as age, disease-stage, treatment, etc. will be explored, and appropriate adjustment will be performed. An economic evaluation will be performed for each randomized group and compared.

ELIGIBILITY:
Inclusion Criteria:

* Lesions suspected for cancer in the colon or rectum recognized through colonoscopy or sigmoidoscopy found at scopy centres in Odense, Nyborg, Svendborg or Slagelse, all in Denmark
* Can speak and understand Danish.

Exclusion Criteria:

* Life-threatening disease: score 4 in the American Society of Anaesthesiologists status classification system.
* Dementia ( Diagnosed or in a diagnostic phase).
* Severe psychiatric disease ( Diagnosed or in a diagnostic phase).
* Mentally retarded ( Diagnosed or in a diagnostic phase).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2016-02-26 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Self evaluated Self Efficacy for Cancer | Change in "Cancer Behaviour Inventory - Brief" from inclusion to measurement 3: one week after receipt of information about treatment end or not later than one year after inclusion.
  Cancer Behaviour Inventory - Brief

SECONDARY OUTCOMES:
Self evaluated Self Efficacy for Cancer | Change in "Cancer Behaviour Inventory - Brief" from inclusion to three days before treatment start.
  Cancer Behaviour Inventory - Brief
Self evaluated Self Efficacy for Cancer | Change in "Cancer Behaviour Inventory - Brief" from inclusion to six weeks after measurement 3.
  Cancer Behaviour Inventory - Brief
Self evaluated Self Efficacy for Cancer | Change in "Cancer Behaviour Inventory - Brief" from three days before treatment start to measurement 3: one week after receipt of information about treatment end or not later than one year after inclusion.
  Cancer Behaviour Inventory - Brief
Self evaluated Self Efficacy for Cancer | Change in "Cancer Behaviour Inventory - Brief" from three days before treatment start to six weeks after measurement 3.
  Cancer Behaviour Inventory - Brief
Self evaluated Self Efficacy for Cancer | Change in "Cancer Behaviour Inventory - Brief" from one week after measurement 3: one week after receipt of information about treatment end or not later than one year after inclusion to six weeks after measure point 3.
  Cancer Behaviour Inventory - Brief
Continuity of care | Change in "Continuity of care" from inclusion to measurement 3: one week after receipt of information about treatment end or not later than one year after inclusion.
  Qualitatively validated questions answered by participants
Continuity of care | Change in "Continuity of care" from inclusion to three days before treatment start.
  Qualitatively validated questions answered by participants
Continuity of care | Change in "Continuity of care" from inclusion to six weeks after measurement 3.
  Qualitatively validated questions answered by participants
Continuity of care | Change in "Continuity of care" from three days before treatment start to measurement 3: one week after receipt of information about treatment end or not later than one year after inclusion.
  Qualitatively validated questions answered by participants
Continuity of care | Change in "Continuity of care" from three days before treatment start to six weeks after measurement 3.
  Qualitatively validated questions answered by participants
Continuity of care | Change in "Continuity of care" from one week after measurement 3: one week after receipt of information about treatment end or not later than one year after inclusion to six weeks after measure point 3.
  Qualitatively validated questions
Unmet needs | Change in "Unmet needs" from three days before treatment start to measurement 3: one week after receipt of information about treatment end or not later than one year after inclusion.
  Patients experienced needs and degree of fulfilled support
Unmet needs | Change in "Unmet needs" from three days before treatment start to six weeks after measurement 3.
  Patients experienced needs and degree of fulfilled support
Unmet needs | Change in "Cancer Behaviour Inventory - Brief" from one week after measurement 3: one week after receipt of information about treatment end or not later than one year after inclusion to six weeks after measure point 3.
  Patients experienced needs and degree of fulfilled support
Health-related Quality of Life | Change in "Health-related Quality of Life" from three days before treatment start to six weeks after measurement 3.
  European Organisation for Research and Treatment of Cancer Quality of life questionnaire with 30 questions (EORCT QLQ-c30).

CONTACTS AND LOCATIONS:
Overall Officials: Lise Fillion, PhD, Study Chair — Nursing Faculty, Laval University; Jens Søndergaard, PhD, Study Chair — Research Unit of General Practice, Faculty of Health Sciences, University of Southern Denmark; Marianne K Thygesen, PhD, Principal Investigator — Surgery department A, Clinical Institute, Faculty of Health Sciences, University of Southern Denmark and OPEN at Region of Southern Denmark; Niels Qvist, DMSc, Study Director — Surgery department A, Clinical Institute, Faculty of Health Sciences, University of Southern Denmark

IPD SHARING:
Plan to Share IPD: No